CLINICAL TRIAL: NCT04123249
Title: Effects of Intravenous Anesthetics vs Inhaled Anesthetics on Early Postoperative Sleep Quality and Complications of Patients After Laparoscopic Surgery Under General Anesthesia
Brief Title: The Effects of Intravenous Anesthetics and Inhaled Anesthetics on Patients' Postoperative Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yanchao Yang (Other)
Responsible Party: Sponsor-Investigator, Yanchao Yang, Principal investigator, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: general anesthetics and sleep
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Sleep Quality; General Anesthesia; Propofol; Sevoflurane; Dreaming
MeSH Terms: interventions — Propofol; Anesthetics, Intravenous; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Propofol (Experimental): In the Group P, propofol 4-6 mg/kg/h and remifentanil 0.2μg/kg/min were infused by intravenous pump separately for assisted sedation and assisted analgesia.
  Interventions: Drug: Propofol
- Group Sevoflurane (Experimental): sevoflurane (concentration: 2%-3%, mixed with 50% air and 50% oxygen to keep the minimum alveolar concentration (MAC) at 1.0-1.1) was inhaled to maintain assisted sedation, and remifentanil 0.2 μg/kg/min was infused by intravenous pump for assisted analgesia.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Group Propofol was given propofol 4mg/kg/h intravenous pumping to assist sedation
  Other Names: Intravenous Anesthetics
  Arms: Group Propofol
Drug: Sevoflurane — Group Sevoflurane was given sevoflurane inhalation maintenance (concentration of 2% to 3% and mixed with 50% oxygen and air) to assist sedation；
  Other Names: Inhaled Anesthetics
  Arms: Group Sevoflurane

SUMMARY:
Adequate sleep is necessary for physical and mental health of human being. Although surgery and anesthesia techniques have improved in resent years, postoperative sleep disturbance remains a challenging problem in surgical procedures1. Postoperative sleep fragmentation and poor sleep quality can not only result in hyperalgesia and a delay in postoperative recovery2, lack of sleep after surgery can also bring many potential adverse effects such as cognitive disorders (such as delusions, delirium), chronic pain, mood disorders, metabolic disorders, and pro-inflammatory changes3-5. Previous studies have reported that age, preoperative comorbidity and severity of surgical trauma were independent factors that associated with postoperative sleep disturbance6,7. Our prior studies have also found that patients are more likely to experience decreased sleep quality after receiving general anesthesia, which was characterized by a decrease in each sleep stage8. Propofol and sevoflurane are commonly used general anesthetics in clinical practice. The choice of anesthetic may also affect the cognitive outcome after surgery, but the results of clinical studies have always been contradictory. Some studies report that the cognitive results after inhalation are worse than those after intravenous anesthesia. And the incidence of dreaming was significantly higher in the sevoflurane anesthesia group compared to the propofol group9-11. Another study conduct among infants proved that compared with propofol-remifentanil, sevoflurane appears to be associated with less sleep disturbances in the first weeks after surgery12. Based on these conflicts, the aim of the current study was to compare the effect of propofol vs sevoflurane on early postoperative sleep quality and complications of patients receiving laparoscopic surgery after general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

ASA : GradeⅠtoⅡ Laparoscopic surgery

Exclusion Criteria:

history of sleep apnea; severe neuropsychiatric disorders; long-term use of sedatives or sleeping pills; can not implement multi-lead sleep monitoring and other sleep disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
postoperative sleep quality of one night before surgery | one night after the surgery
  Use sleep monitor to test the sleep quality one night before surgery
postoperative sleep quality of the first night after surgery | the first night after surgery
  Use sleep monitor to test the sleep quality the first night after surgery
postoperative sleep quality of the third night after surgery | the third night after surgery
  Use sleep monitor to test the sleep quality the third night after surgery

SECONDARY OUTCOMES:
Postoperative pain score | 24h after surgery
  Use visual analog scale (VAS) score, where 0 means no pain and 10 means severe pain,to evaluate pain scores after surgery
postoperative adverse effect | 24 hours after surgery
  record the adverse reactions such as respiratory depression, bradycardia, nausea, vomiting and dizziness within 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China